CLINICAL TRIAL: NCT03804021
Title: Post-treatment Long-term Follow-up Study of ADVM-043 Gene Therapy in Alpha-1 Antitrypsin Deficiency
Brief Title: Long-Term Follow-up Study of ADVM-043
Status: Completed | Type: Observational
Sponsor: Adverum Biotechnologies, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ADVM-043-03
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Results first posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2023-09

CONDITIONS: Alpha-1 Antitrypsin Deficiency
Keywords: Alpha-1 Antitrypsin Deficiency; alpha1-antitrypsin deficiency; alpha 1-antitrypsin deficiency; alpha1AT; A1AT; ADVM-043; AAVrh.10halpha1AT; AAVrh.10hA1AT; Gene transfer vector; Gene therapy; Lung disease; Emphysema; COPD; ADVANCE study; Long Term Follow Up
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Lung Diseases; Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Roll over: Subjects who received ADVM-043 in a parent study (ADVANCE; NCT02168686)
  Interventions: Genetic: No Intervention

INTERVENTIONS:
Genetic: No Intervention — Subjects who received ADVM-043 in a parent study (ADVANCE; NCT02168686)

SUMMARY:
ADVM-043-03 is a long-term follow-up (LTFU) study of subjects who participated in the ADVM-043-01 (NCT02168686) multi-center gene therapy clinical study (ADVANCE) that evaluated ADVM-043 for the treatment of Alpha-1 Antitrypsin (A1AT) deficiency.

DETAILED DESCRIPTION:
ADVM-043-03 was a multi-center, observational study without administration of the ADVM-043 investigational product. Subjects who participated in the ADVANCE study (ADVM-043-01; NCT02168686) were enrolled into this LTFU study for continued safety monitoring for a 2-year period.

ELIGIBILITY:
Key Inclusion Criteria:

* The subject has A1AT deficiency and has previously received ADVM-043 gene therapy

Key Exclusion Criteria:

* The subject is unwilling or unable to participate in all required study evaluations in the long-term follow-up protocol
* The subject is participating in another investigational treatment protocol
* The subject is unable to understand the purpose and risks of the study or cannot provide a signed and dated informed consent form (ICF)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who received ADVM-043 in a treatment protocol
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2018-12-27 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2021-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charlton Strange, MD, Principal Investigator — Medical University of South Carolina, Charleston, SC, USA; Mark Brantly, MD, Principal Investigator — University of Florida, Gainesville, FL, USA
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - Medical University of South Carolina, Charleston, South Carolina

REFERENCES:
- [Derived] Remih K, Amzou S, Strnad P. Alpha1-antitrypsin deficiency: New therapies on the horizon. Curr Opin Pharmacol. 2021 Aug;59:149-156. doi: 10.1016/j.coph.2021.06.001. Epub 2021 Jul 10. PMID 34256305

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a long-term follow-up study for subjects who previously participated in Study ADVM-043-01.
Pre-assignment Details: Completion of Study ADVM-043-01
Groups:
- Study ADVM-043-01 Part A Dose Level 1: Single IV infusion of ADVM-043 at 8E13 total vg
- Study ADVM-043-01 Part A Dose Level 2: Single IV infusion of ADVM-043 at 4E14 total vg
- Study ADVM-043-01 Part A Dose Level 3: Single IV infusion of ADVM-043 at 1.2E15 total vg
Period: Overall Study
Arm/Group | Study ADVM-043-01 Part A Dose Level 1 | Study ADVM-043-01 Part A Dose Level 2 | Study ADVM-043-01 Part A Dose Level 3
Started | 2 | 2 | 2
Completed | 2 | 2 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: [Not Specified]
Groups:
- Total: Total of all reporting groups
Arm/Group | Study ADVM-043-01 Part A Dose Level 1 | Study ADVM-043-01 Part A Dose Level 2 | Study ADVM-043-01 Part A Dose Level 3 | Total
Number analyzed (Participants) | 2 | 2 | 2 | 6
Age, Continuous [Mean (Full Range); unit: years] | 40.5 [25 to 56] | 53.5 [52 to 55] | 61.0 [53 to 69] | 51.7 [25 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 3
  Male | 2 | 1 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 2 | 2 | 6
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events of Special Interest and of Serious Adverse Events Related to ADVM-043
Description: All adverse events of special interest and all serious adverse events related to ADVM-043
Time Frame: 2 years from start of long-term follow-up study ADVM-043-03 (NCT03804021) (2 years from completion of the parent study (ADVM-043-01, NCT02168686)
Population: Subjects who received ADVM-043 in Study ADVM-043-01
Measure: Number; unit: participants
Groups:
- Study ADVM-043-01 Part A Dose Level 1: Follow-up after single IV infusion of ADVM-043 8E13 total vg
- Study ADVM-043-01 Part A Dose Level 2: Follow-up after single IV infusion of ADVM-043 4E14 total vg
- Study ADVM-043-01 Part A Dose Level 3: Follow-up after single IV infusion of ADVM-043 1.2E15 total vg
Arm/Group | Study ADVM-043-01 Part A Dose Level 1 | Study ADVM-043-01 Part A Dose Level 2 | Study ADVM-043-01 Part A Dose Level 3
Number analyzed (Participants) | 2 | 2 | 2
participants
  Deaths | 0 | 0 | 0
  Serious Adverse Events | 0 | 0 | 0
  Other Adverse Events | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years from start of long-term follow-up study ADVM-043-03 (NCT03804021) (2 years from completion of the parent study (ADVM-043-01, NCT02168686)
Description: All adverse events of special interest and all serious adverse events related to ADVM-043
Arm/Group | Study ADVM-043-01 Part A Dose Level 1 | Study ADVM-043-01 Part A Dose Level 2 | Study ADVM-043-01 Part A Dose Level 3
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 1/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure restrictions on the PIs are that Sponsor can review communications by the PI prior to public release and can embargo communications regarding trial results for varying time periods from the time submitted to the sponsor for review. The Sponsor may require changes to the communication after review and may delay publication upon request by the Sponsor to allow the Sponsor to seek/obtain patent protection.

DOCUMENTS (2):
  • Study Protocol (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/21/NCT03804021/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-02): https://cdn.clinicaltrials.gov/large-docs/21/NCT03804021/SAP_001.pdf